CLINICAL TRIAL: NCT04609007
Title: The Effect of a Brief Intervention for Problem Gamblers - a Randomized Controlled
Brief Title: The Effect of a Brief Intervention for Problem Gamblers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Clara Hellner Gumpert, Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017/1063-31
Record Dates: First submitted 2018-08-30; First posted 2020-10-30 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Gambling Problem
MeSH Terms: interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as usual (Active Comparator): The TAU condition consists of a single session of regular help-line telephone counselling
  Interventions: Behavioral: Regular help-line telephone counselling
- Cognitive behavioral therapy (Experimental): The experimental condition consists of a single session of regular help-line telephone counselling plus four therapist guided online CBT sessions.
  Interventions: Behavioral: Cognitive behavioral therapy (CBT)

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy (CBT) — A brief 4 sessions online CBT program with therapist support.
  Arms: Cognitive behavioral therapy
Behavioral: Regular help-line telephone counselling — A single session of telephone counselling with a help-line counsellor
  Arms: Treatment as usual

SUMMARY:
A pragmatic randomized pilot trial primarily examining the feasibility of a brief therapist guided online self-help program based on Cognitive behavioral therapy (CBT). Participants will be randomized to either a treatment as usual condition (TAU) or to TAU plus CBT.

DETAILED DESCRIPTION:
The current study is a pragmatic randomized pilot trial examining the feasibility and effects of a brief therapist guided online self-help program based on Cognitive behavioral therapy (CBT) . Participants will be randomized to either a treatment as usual condition (TAU) or to TAU plus CBT.

Participants will be recruited via the Swedish national gambling helpline. After assessment for eligibility participants will be randomized, using block randomization to ensure balanced groups, to either TAU or TAU+CBT.

The participants will be measured; at baseline, weekly during the intervention (6 weeks), immediately after the intervention and at 6 weeks after treatment termination. Informed consent will be collected prior any data collection.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years
* Experiencing gambling problems (PGSI ≥ 3 p)
* Good enough knowledge in Swedish
* Access to a smart phone or computer with internet connection

Exclusion Criteria:

* Being involved in another treatment study the previous 3 months
* Other concurrent treatment for gambling problems
* Being on a non-stable pharmacological treatment for any psychiatric condition
* Severe depression defined as a PHQ-9 score of 20 points or more

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Retention at the end of the study | 6-weeks after the intervention
  Retention, defined as proportion of participants who fill out the last follow-up survey
Time for execution of the study | from the date of the first included participant to the last included, assessed up to 52 weeks
  Time for execution of the study as measured by the time from the first included participant to the last included,
Participant rated satisfaction with the treatment protocol | measured in conjunction with each online treatment module for up to six weeks (at four occasions)
  Participant rated satisfaction with the treatment protocol will be measured using three items at the end of each online treatment module. The items are measured on a VAS scale ranging from 1-5 (1= not at all, 5 = very).
  Item 1) "How helpful do you think the content of this module has been?" Item 2) "How well does the content of the module fit the problems you experience and want help with?" Item 3) "What grade from 1 to 5 would you give this module?
Participant rated satisfaction with the treatment at large | immediately after the intervention.
  Participant rated satisfaction with the treatment at large will be measured immediately after the intervention using 12 items on a VAS scale ranging from 1 (not at all) to 10 (very). Item 8 answers "yes" or "no" and item 9 is a free-text entry only available if item 8 answers "yes". Items 1- 4 and items 10-12 captures satisfaction with the program and items 5 - 9 captures satisfaction with the therapist.

SECONDARY OUTCOMES:
Timeline follow-back, days gambling and net losses due to gambling | At baseline, weekly during the intervention, immediately after the intervention and at the 6-weeks follow-up
  A calendar function where gamblers registers days gambling and nett losses due to gambling.
Problem Gambling Severity Index (PGSI) | At baseline and at the 6-weeks follow-up
  An instrument measuring level of gambling problems using 9 items on a 4 levels Likert-scale, 0 p (never) to 3 p (always), with a total score ranging from 0 to 27 p. Scoring 5 points or more indicates problem gambling.
National Opinion Research Center Diagnostic and Statistical Manual of Mental Disorders-IV Screen for Gambling (NODS) | At baseline, immediately after the intervention and at the 6-weeks follow-up
  An instrument measuring measuring gambling disorder. The instrument consists of 17 items which are market "yes" or "no" and yields a total score of 10 points. Five points or more indicates a pathological gambler.
Alcohol Use Disorders Identification Consumption (AUDIT-C) | At baseline, immediately after the intervention and at the 6-weeks follow-up
  An instrument which measures alcohol consumption in the general population. The instrument consists of 3 questions ranging from 0 to 4 with a total score of 0-12 points. A total score of ≥ 6 p indicates alcohol problems in men and ≥ 4 p in women
Drug Use Disorders Identification Test Consumption (DUDIT-C) | At baseline, immediately after the intervention and at the 6-weeks follow-up
  An instrument consisting of 3 items measuring illicit drug consumption.
Generalised Anxiety Disorder 7-item scale (GAD-7) | At baseline, immediately after the intervention and at the 6-weeks follow-up
  An instrument measuring anxiety consisting of 7 items with a total score ranging from 0 to 21 points where 15 or more points indicates severe anxiety.
Gambling Abstinence Self-Efficacy Scale (GASS) | At baseline, immediately after the intervention and at the 6-weeks follow-up
  An instrument measuring self efficacy in gambling situations. The instrument consists of 21 items scored 0 to 5 points, yielding a total score of 0 - 105 points.
Gambling Urges Scale (GUS) | At baseline, immediately after the intervention and at the 6-weeks follow-up
  An instrument measuring gambling urges. The instrument consists of 6 items on a Likert-scale 0 to 7, yielding a total score ranging from 0 - 42 points. A higher total score indicates more gambling urges.
Consumption Screen for Problematic Gambling (CSPG) | At baseline
  An instrument measuring consumption of gambling the previous year. The instrument consists of three items yielding a total score ranging from 0-13 points. Four or more points indicates gambling problems
Patient Health Questionnaire-9 (PHQ-9) | At baseline, immediately after the intervention and at the 6-weeks follow-up
  A nine items instrument measuring depression ranging from 0 to 27 points. Twenty points or more indicates severe depression
World Health Organization Quality of Life Instruments (WHOQOL-BREF) | At baseline, immediately after the intervention and at the 6-weeks follow-up
  A 26 items instrument developed by the World Health Organisation measuring quality of life. Items are scored 1-5 points, yielding a total score ranging from 26 - 130 p.

CONTACTS AND LOCATIONS:
Overall Officials: Clara Hellner, Professor, Principal Investigator — Karolinska Institutet
Locations (1):
- Stockholm Center for Psychiatry Research, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wall H, Magnusson K, Hellner C, Andersson G, Jayaram-Lindstrom N, Rosendahl I. The evaluation of a brief ICBT program with therapist support for individuals with gambling problems in the context of a gambling helpline: a randomized pilot trial. Pilot Feasibility Stud. 2023 Feb 17;9(1):26. doi: 10.1186/s40814-023-01257-7. PMID 36805024

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-06): https://cdn.clinicaltrials.gov/large-docs/07/NCT04609007/Prot_SAP_000.pdf